CLINICAL TRIAL: NCT05439811
Title: Retrospective Data Analysis on the Application of Swan-Ganz Catheter in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Shanglong Yao, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: SGCS
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Complications
Keywords: Swan-Ganz Catheter; Cardiac Surgery; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Swan-Ganz Catheter — Swan-Ganz Catheter

SUMMARY:
The investigators aimed to investigate postoperative complications associated with Swan-Ganz Catheter based on the clinical data of Wuhan Union Hospital and Wuhan Asian heart hospital for 10 years, including major cardiovascular, respiratory adverse events, ICU time, mechanical ventilation time, length of hospital stay, in-hospital mortality, and 30-day postoperative mortality events.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Patients undergoing major cardiac surgery under general anesthesia;
* Patients with complete sex, age, use of floating catheter and prognosis data

Exclusion Criteria:

* ASA grade V and above;
* End stage renal disease requiring (or undergoing) renal replacement therapy;
* Pregnant or lactating women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cardiovascular events | one week after operation
  1) Cardiac death; 2) Non fatal myocardial infarction; 3) Intra aortic balloon counterpulsation (IABP); 4) Thoracotomy exploration; 5) Heart failure.
Number of participants respiratory adverse events | one week after operation
  1) Acute lung injury: Diagnosis according to Berlin diagnostic standard; 2) Atelectasis: X-ray confirmed with body temperature >37.5c or abnormal pulmonary manifestations; 3) Pneumothorax: chest X-ray diagnosis; 4) Pneumonia: confirmed by radiology or bacteriology

IPD SHARING:
Plan to Share IPD: Undecided
If the patient's privacy information is not involved, you can contact the research team by email to obtain data (yaoshanglong@hust.edu.cn)